CLINICAL TRIAL: NCT04591717
Title: Phase 1b Open-Label Study of the Safety, Reactogenicity, and Immunogenicity of Prophylactic Vaccination With 2nd Generation (E1/E2B/E3-Deleted) Adenoviral-COVID-19 in Normal Healthy Volunteers
Brief Title: COVID-19 Vaccination Using a 2nd Generation (E1/E2B/E3-Deleted) Adenoviral-COVID-19 in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-COVID-19-hAd5-Vaccine
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: 0.5 mL of hAd5-S-Fusion+N-ETSD SC (Experimental): 0.5 mL of hAd5-S-Fusion+N-ETSD SC (5 × 10e10 VP/dose) on days 1 and 22
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 2: 1.0 mL of hAd5-S-Fusion+N-ETSD SC (Experimental): Cohort 2: 1.0 mL of hAd5-S-Fusion+N-ETSD SC (1 × 10e11 VP/dose) on days 1 and 22
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 3a: 1.0 mL of hAd5-S-Fusion+N-ETSD SC and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (Experimental): Cohort 3a: 1.0 mL of hAd5-S-Fusion+N-ETSD SC (1 × 10e11 VP/dose) and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (5 × 10e10 VP/dose) on day 1; 1.0 mL of hAd5-S-Fusion+N-ETSD SC (1 × 10e11 VP/dose) and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (5 × 10e10 VP/dose) on day 22
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 3b: 1.0 mL of hAd5-S-Fusion+N-ETSD SC and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (Experimental): Cohort 3b: 1.0 mL of hAd5-S-Fusion+N-ETSD SC (1 × 10e11 VP/dose) and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (5 × 10e10 VP/dose) on day 1; no vaccine on day 22
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 3c: 1.0 mL of hAd5-S-Fusion+N-ETSD SC and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (Experimental): Cohort 3c: 1.0 mL of hAd5-S-Fusion+N-ETSD SC (1 × 10e11 VP/dose) and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (5 × 10e10 VP/dose) on day 1; 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (5 × 10e10 VP/dose) on day 22
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 3d: 1.0 mL of hAd5-S-Fusion+N-ETSD SC and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (Experimental): Cohort 3d: 1.0 mL of hAd5-S-Fusion+N-ETSD SC (1 × 10e11 VP/dose) and 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (5 × 10e10 VP/dose) on day 1; 0.5 mL of hAd5-S-Fusion+N-ETSD sublingually (5 × 10e10 VP/dose) on days 15 and 29
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine

INTERVENTIONS:
Biological: hAd5-S-Fusion+N-ETSD vaccine — The hAd5-S-Fusion+N-ETSD Vaccine is a human adenovirus serotype 5 (hAd5) vector with E1/E2b/E3 deletions expressing SARS-CoV-2 viral antigen spike fusion protein and nucleocapsid with an enhanced T-cell stimulation domain.

SUMMARY:
This is a phase 1b, open-label study in adult healthy subjects. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of the hAd5-S-Fusion+N-ETSD vaccine and select a dose for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, age 18 - 55 years, inclusive, at time of enrollment.
2. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
3. Agrees to the collection of biospecimens (eg, nasopharyngeal [NP] swabs) and venous blood per protocol.
4. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
5. Temperature < 38°C.
6. Negative for SARS-CoV-2 (qPCR or LAMP test) and no known previous COVID-19 exposure or disease.
7. Agreement to practice effective contraception for female subjects of childbearing

potential and non-sterile males. Female subjects of childbearing potential must agree to use effective contraception while on study until at least 1 month after the last dose of vaccine. Non-sterile male subjects must agree to use a condom while on study until at least 1 month after the last dose of vaccine. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), oral contraceptives, and abstinence.

Exclusion Criteria:

1. Allergy to any component of the investigational vaccine, or a more severe allergic reaction and history of allergies in the past.
2. Pregnant and nursing women. A negative serum or urine pregnancy test during screening and on the day of and prior to each dose must be documented before the vaccine is administered to a female subject of childbearing potential.
3. Live in a nursing home or long-term care facility.
4. Chronic lung disease including chronic obstructive pulmonary disease (COPD) or moderate to severe asthma.
5. Pulmonary fibrosis.
6. Active smoker.
7. Bone marrow or organ transplantation.
8. Obesity (defined as body mass index [BMI] of 30 kg/m2 or higher).
9. Diabetes.
10. Chronic kidney disease.
11. Liver disease.
12. Sickle cell disease.
13. Thalassemia.
14. Doctors, nurses, first responders, and other healthcare workers working in direct contact with COVID-19 patients.
15. Any disease associated with acute fever, or any infection.
16. Self-reported history of severe acute respiratory syndrome (SARS).
17. History of hepatitis B or hepatitis C.
18. HIV or other acquired or hereditary immunodeficiency.
19. Serious cardiovascular diseases, such as heart failure, coronary artery disease, cardiomyopathies, arrhythmia, conduction block, myocardial infarction, pulmonary hypertension, severe hypertension without controllable drugs, etc.
20. Cerebrovascular disease.
21. Cystic fibrosis.
22. Neurologic conditions, such as dementia.
23. Hereditary or acquired angioneurotic edema.
24. Urticaria in the last 12 months.
25. No spleen or functional asplenia.
26. Platelet disorder or other bleeding disorder that may cause injection contraindication.
27. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness within 3 months before administration of study vaccine. (Including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators. The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.)
28. Prior administration of blood products in last 4 months.
29. Prior administration of other research medicines in last 1 month.
30. Received or plans to receive an attenuated vaccine within 1 month before or after each study vaccination.
31. Received or plans to receive an inactivated vaccine within 14 days before or after each study vaccination.
32. Current treatment with investigational agents for prophylaxis of COVID-19.
33. Have a household contact that has been diagnosed with COVID-19.
34. Current anti-tuberculosis prophylaxis or therapy.
35. Currently receiving treatment for cancer or history of cancer in the last five years (except basal cell carcinoma of the skin and cervical carcinoma in situ).
36. According to the judgement of investigator, various medical, psychological, social or other conditions that could affect the subjects ability to sign informed consent.
37. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Incidence of MAAEs and SAEs | 1 week
  Incidence of MAAEs and SAEs through 1 week post final vaccine administration
Incidence and severity of solicited local reactogenicity AEs | 1 week
  Incidence and severity of solicited local reactogenicity AEs through 1 week post final vaccine administration
Incidence and severity of solicited systemic reactogenicity AEs | 1 week
  Incidence and severity of solicited systemic reactogenicity AEs through 1 week post final vaccine administration
Incidence and severity of unsolicited AEs | 1 week
  Incidence and severity of unsolicited AEs through 1 week post final vaccine administration
Incidence of MAAEs and SAEs | 30 days to 6 months
  Incidence of MAAEs and SAEs through 30 days and 6 months post final vaccine administration
Incidence and severity of unsolicited AEs | 30 days
  Incidence and severity of unsolicited AEs through 30 days post final vaccine administration
Incidence of abnormal changes of laboratory safety examinations | 30 days
  Incidence of abnormal changes of laboratory safety examinations
Vital Signs - Fever | 30 days
  Changes in vital signs from Grades 1-4:
  - Fever - measured in (°C) or (°F)
Vital Signs - Tachycardia | 30 Days
  Changes in vital signs from Grades 1-4:
  - Tachycardia - measured in beats per minute
Vital Signs - Bradycardia | 30 Days
  Changes in vital signs from Grades 1-4:
  - Bradycardia - measured in how many beats per minute
Vital Signs - Hypertension | 30 Days
  Changes in vital signs from Grades 1-4:
  - Hypertension (systolic/diastolic) - measured in mm Hg
Vital Signs - Hypotension | 30 Days
  Changes in vital signs from Grades 1-4:
  - Hypotension (systolic) - measured in mm Hg
Vital Signs - Respiratory Rate | 30 Days
  Changes in vital signs from Grades 1-4:
  - Respiratory Rate - measured in how many breaths per minute
GMFR in IgG titer | Day 387
  GMFR in IgG titer
GMT of S-specific, RBD-specific, and N-specific antibodies against 2019 novel coronavirus | Day 387
  GMT of S-specific, RBD-specific, and N-specific antibodies against 2019 novel coronavirus tested by ELISA in serum
Percentage of subjects who seroconverted | Day 387
  Percentage of subjects who seroconverted (as defined as 4-fold change in antibody titer relative to baseline)
GMFR in neutralizing antibody | Day 387
  GMFR in neutralizing antibody
GMT | Day 387
  GMT of neutralizing antibody
Seroconversion rate of neutralizing antibody | Day 387
  Seroconversion rate of neutralizing antibody (as defined as 4-fold change in antibody titer relative to baseline)
CD8+ T-Cell activity against SARS-CoV-2 S protein, RBD, and N protein | Day 387
  CD8+ T-Cell activity against SARS-CoV-2 S protein, RBD, and N protein measured by ELISPOT assay
CD4+ T-Cell activity against SARS-CoV-2 S protein, RBD, and N protein | Day 387
  CD4+ T-Cell activity against SARS-CoV-2 S protein, RBD, and N protein measured by standard immune assay

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chan Soon - Shiong Institute for Medicine, El Segundo, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California

IPD SHARING:
Plan to Share IPD: No